CLINICAL TRIAL: NCT01570816
Title: Improving Ambulatory Community Access After Paralysis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rudi Kobetic, Biomedical Engineer, Louis Stokes VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12004-H02; 1I01RX000528-01A2 (NIH)
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Stroke; Partial Paralysis; Spinal Cord Injury; Tetraplegia; Quadriplegia
Keywords: stroke; partial paralysis; gait correction; functional electrical stimulation; paraplegia; tetraplegia; spinal cord injury
MeSH Terms: conditions — Stroke; Muscle Weakness; Spinal Cord Injuries; Quadriplegia; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Volunteers are evaluated for appropriateness for inclusion in the study on an intent-to-treat basis. Qualifying candidates all receive the implanted neuroprosthesis and participate in post-operative training and follow-up procedures
  Interventions: Device: IRS-8 (8 channel implanted receiver stimulator)

INTERVENTIONS:
Device: IRS-8 (8 channel implanted receiver stimulator) — Surgical implantation of an 8 channel pulse generator to stimulate paralyzed muscles of the lower extremities
  Other Names: Implanted pulse generator for ambulation; Implanted FES system for lower extremities; Implated FES system for ambulation; FES system for walking; Implanted neuroprosthesis for gait correction; Gait correction in partial paralysis

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of functional electrical stimulation (FES) provided by an implanted pulse generator (IPG) in correcting hip, knee and ankle function to improve walking in people with partial paralysis.

DETAILED DESCRIPTION:
In a surgical procedure electrodes are inserted into muscles of the lower extremities to correct hip, knee and ankle function. The electrode leads are connected to an implanted pulse generator located in the abdomen. After a typical post-operative period of two to five days, the recipient will be discharged home for two to six weeks of moderate activity. Following a 6 week period of laboratory exercise and training, functional use of the neuroprosthesis will begin at home and in the community with follow-up evaluations at 1, 3, 6 and 12 months. Laboratory assessments include walking speed and distance, physiologic cost, muscle strength, measure of spasticity, and gait analysis with and without stimulation. A number of self-reporting instruments are administered to capture individual's participation, quality of life and various aspects of perceived community ambulation.

ELIGIBILITY:
Inclusion Criteria:

* problems walking because of paralysis for more than 6 months
* weak hip flexors and extensors or excessive tone
* weak ankle dorsiflexors (muscles bringing the foot up)
* weak plantar flexors (ankle muscles for push-off)
* foot drop that is causing "dragging" or "catching" toes during walking
* swinging the leg sideways or hiking the hip to clear affected leg during stepping
* endurance to walk at least 10 ft with minimal assistance
* hip extension range to neutral
* hip flexion range greater or equal to 90 degrees
* ankle range to neutral
* sufficient upper extremity function to use a walking aid
* muscles respond to electrical stimulation

Exclusion Criteria:

* cardiac arrythmias
* demand pacemaker
* pregnancy
* Parkinson's disease
* traumatic brain injury
* autoimmune deficiency
* uncontrolled diabetes
* significant edema of the affected limb
* active pressure ulcers or open wounds
* sepsis or an active infection
* severe osteoporosis
* uncontrolled seizures
* moderate depression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2012-04; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
The effect of functional electrical stimulation of the hip, knee and ankle muscles to improve walking in people with partial paralysis | up to 36 months
  Experiments involving analyses of individual's speed, distance and quality of walking will be performed both with and without stimulation to determine if individuals are able to improve community ambulatory access with use of neuroprosthesis.

SECONDARY OUTCOMES:
Feasibility of initiating a step with a trigger from an accelerometer incorporated in the external control unit to adjust to environmental circumstances and situations encountered in community ambulation | up to 36 months
  Experiments involving analyses of individual's speed, distance and quality of walking will be performed both with and without accelerometer triggered stepping to determine if individuals are able to adjust to environmental circumstances and situations encountered in community ambulation.

CONTACTS AND LOCATIONS:
Overall Officials: Rudi Kobetic, MSBE, Principal Investigator — Louis Stokes Cleveland Dept. of Veterans Affairs Medical Center
Locations (1):
- Louis Stokes Cleveland Dept. of Veterans Affairs Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Bailey SN, Hardin EC, Kobetic R, Boggs LM, Pinault G, Triolo RJ. Neurotherapeutic and neuroprosthetic effects of implanted functional electrical stimulation for ambulation after incomplete spinal cord injury. J Rehabil Res Dev. 2010;47(1):7-16. doi: 10.1682/jrrd.2009.03.0034. PMID 20437323
- [Background] Hardin E, Kobetic R, Murray L, Corado-Ahmed M, Pinault G, Sakai J, Bailey SN, Ho C, Triolo RJ. Walking after incomplete spinal cord injury using an implanted FES system: a case report. J Rehabil Res Dev. 2007;44(3):333-46. doi: 10.1682/jrrd.2007.03.0333. PMID 18247230
- [Derived] Triolo RJ, Bailey SN, Foglyano KM, Kobetic R, Lombardo LM, Miller ME, Pinault G. Long-Term Performance and User Satisfaction With Implanted Neuroprostheses for Upright Mobility After Paraplegia: 2- to 14-Year Follow-Up. Arch Phys Med Rehabil. 2018 Feb;99(2):289-298. doi: 10.1016/j.apmr.2017.08.470. Epub 2017 Sep 9. PMID 28899825
- See also: Cleveland FES center website — http://fescenter.org